CLINICAL TRIAL: NCT05746546
Title: Open Label Extension Study of Depressed Mood Improvement Through Nicotine (Depressed MIND3)
Brief Title: Depressed Mood Improvement Through Nicotine Dosing-3 (Depressed MIND3) Extension
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Warren Taylor, Professor of Psychiatry, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 222009-EXT; 4R33MH122464-03 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-02-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Depressive Disorder
Keywords: Geriatrics; aging; elderly; cognition; memory; Transdermal Nicotine Patch; depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transdermal Nicotine Patch (Experimental): Participants will wear nicotine transdermal patches daily for 12-15 weeks. Participants will apply a study patch each morning and remove at bedtime. Active dose will titrate up from 3.5mg to 7mg, and then can optionally be further titrated to a maximum dose of 14mg. After week12, the dose will be slowly tapered over 2-3 weeks.
  Interventions: Drug: Transdermal Nicotine patch

INTERVENTIONS:
Drug: Transdermal Nicotine patch — Participants will wear nicotine transdermal patches daily for 12-15 weeks. Participants will apply a study patch each morning and remove at bedtime. Active dose will titrate up from 3.5mg to 7mg, and then can optionally be further titrated to a maximum dose of 14mg. After week12, the dose will be slowly tapered over 2-3 weeks.
  Other Names: Nicoderm CQ; Nicotrol

SUMMARY:
Deficits in cognitive control are core features of late-life depression (LLD), contributing both to emotion dysregulation and problems with inhibiting irrelevant information, conflict detection, and working memory. Clinically characterized as executive dysfunction, these deficits are associated with poor response to antidepressants and higher levels of disability. Improvement of cognitive control network (CCN) dysfunction may benefit both mood and cognitive performance, however no current pharmacotherapy improves Cognitive Control Network deficits in LLD.

The study examines the hypothesis that nicotine acetylcholine receptor agonists enhance Cognitive Control Network function. This effect may resultantly improve mood and cognitive performance in LLD. Small, open-label studies of transdermal nicotine (TDN) patches have supported potential clinical benefit and provided support that transdermal nicotine administration engages the Cognitive Control Network.

This is an open-label, extension to the blinded Depressed MIND 3 (Depressed Mood Improvement through nicotine dosing) study. It will evaluate longer-term safety and efficacy of Transdermal Nicotine Patches for potential benefit in cognitive and depression outcomes in elderly depressed participants. Subjects complete blinded randomized trial of Depressed MIND-3 will be eligible for continuation in this extension. This extension study will consist of up to 12 weeks of treatment and a 3 -week safety follow-up period.

DETAILED DESCRIPTION:
The purpose of this open-label extension to the Depressed MIND 3 study will be to gather data on longer-term benefits and safety in patients with late-life depression (LLD). Neuronal nicotinic receptors have long been known to play a critical role in memory function in preclinical studies, with nicotine improving attention, learning, and memory function. This may be particularly relevant in LLD, which is characterized both by affective symptoms and broad cognitive deficits. The co-occurrence of cognitive deficits in LLD is a clinically relevant phenotype characterized by significant disability and poor antidepressant response. Cognitive deficits can persist even with successful antidepressant treatment and increase the risk of depression relapse. Despite the clinical importance of cognitive deficits in LLD, there are no established treatments that specifically target cognition in this population. The lack of clear pharmacologic targets and therapies aimed at improving cognitive deficits in depression is a substantial deficiency in current therapeutics.

Investigators propose that modulation of the cognitive control network by stimulation of cholinergic system nicotinic acetylcholine receptors will improve both mood and cognition in depressed elders. The study is an open-label extension of a randomized double blind placebo control trial that will enroll 80 participants over a 3-year period. After randomization and completion of the blinded study phase, participants will be eligible for this 12-week extension.

At the completion of Week-12 visit of the Depressed MIND -3, all eligible subjects will be offered enrollment in the open label extension study. Study visits during the treatment period for all subjects will occur approximately 3 weeks with flexible dose titration. This will be followed by a 1-3 week taper phase. The total duration of study participation will be approximately 15 weeks.

ELIGIBILITY:
Only individuals who complete 12 weeks of the blinded Depressed MIND trial will be eligible for enrollment.

Eligibility criteria for the blinded phase includes:

Inclusion Criteria:

1. Age ≥ 60 years;
2. Diagnosis of major depressive disorder, single or recurrent episode (DSM5);
3. On a stable therapeutic dose of an allowed SSRI or SNRI for at least 8 weeks;
4. Severity: Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 15;
5. Cognition: Mini-Mental State Examination (MMSE) score ≥ 24;
6. Fluent in English

Exclusion Criteria:

1. Other Axis I psychiatric disorders, except for generalized anxiety disorder (GAD) or social phobia symptoms occurring in a depressive episode or diagnosis of an attentional disorder, such as Attention Deficit Hyperactivity Disorder (ADHD);
2. Use of other augmentation medication treatments for depression, or ADHD e.g., stimulant medications,, e.g., adjunctive bupropion or other augmenting agents, that the participant does not want to stop, although short-acting sedatives are allowed (see below);
3. Any use of tobacco or nicotine in the last year;
4. Living with a smoker or regular exposure to secondhand smoke;
5. History of alcohol use disorder or substance use disorder of moderate or greater severity (endorsing 4 or more of the 12 criteria) in the last 12 months;
6. Acute suicidality;
7. Acute grief (<1 month);
8. Current or past psychosis;
9. Primary neurological disorder, including dementia, stroke, epilepsy, etc.;
10. MRI contraindication;
11. Electroconvulsive therapy or transcranial magnetic stimulation in last 2 months;
12. Current or planned psychotherapy;
13. Allergy or hypersensitivity to nicotine patches;
14. In the last 4 weeks, regular use of drugs with central cholinergic or anticholinergic properties or moderate / severe CYP2A6 inhibitors /inducers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS (Montgomery Asberg Depression Rating Scale) Score | Baseline to week 12
  Primary mood outcome measured by the total score of the clinician rated MADRS. MADRS will be measured every 3 weeks (baseline, week 3, week 6, week 9, and week 12). MADRS total score range is 0-60, where higher scores indicate greater depression severity.
Change in Continuous Performance Task (CPT) Performance | Baseline to Week 12
  Primary cognitive outcome, the CPT is a neuropsychological test that is conducted as part of the NIH EXAMINER Test Battery. Participants are asked to respond to a target image, and not to other images. This test is conducted at baseline and at week12. The specific primary outcome metric is standard error of change in the inter-stimulus hit reaction time or variability between different trials. There is not absolute range, but lower scores indicate decreased variability across trials and overall better performance.

SECONDARY OUTCOMES:
NIH EXAMINER Test Battery | Baseline to Week 12
  Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. We will examine its Executive Composite Score and the three factor scores (Cognitive Control, Fluency, and Working Memory). Higher scores indicate better performance.
Selective Reminding Task | Baseline to Week 12
  Secondary cognitive outcome, Selective Reminding Task as a test of immediate and delayed verbal memory. This is an 8-trial, 16-word test where the interviewer reads unrelated words to the participant who must recall them. Any missed items are then repeated before the next attempt. Alternative word lists are available for repeated assessments. A delayed trial is administered after 20 minutes. Change in the recall, failure to recall and consistency over 12 weeks reflect the verbal memory function.
Trait Adjectives Task | Baseline to Week 12
  Participants view a series of randomized, rapidly presented positive and negative characteristics and quickly indicate whether each adjective does or does not apply to them. Positive and negative adjectives are balanced. Measures include number of adjectives endorsed or rejected, and RT for those trials. Task performance assesses self-referential negativity bias and is associated with antidepressant response. Anticipate increased endorsement of positive adjective and increased rejection of negative adjectives in the active arm.
Ruminative Response Scale | Baseline to Week 12
  Secondary mood outcome: Change in rumination measured by the Ruminative Response Scale total score measured at Screening visit, week 6 and week 12. This is a self-report scale with a range of 0-66, where higher scores indicate higher levels of rumination.
Apathy Evaluation Scale (AES) | Baseline to Week 12
  Secondary Mood Outcomes: Change in apathy as measured by the self-report AES, a questionnaire with a range of 0-54, where lower scores indicate greater apathy.
Insomnia Severity Index | Baseline to Week 12
  Secondary Mood Outcomes: Change in the severity of insomnia measures as self-report, a questionnaire with the range of 0-21, where higher scores indicate increase in severity.
Penn State Worry Questionnaire (PSWQ | Baseline to Week 12
  Secondary mood outcome: Change in anxiety and worry measured by PSWQ, a self-report questionnaire with a range of 16-80, where higher scores indicate greater anxiety and worry.
Fatigue Severity Scale | Baseline to Week 12
  Secondary fatigue out come :self-reported questionnaire that ranges from 0- 56;where higher scores indicate severe fatigue.
General Anxiety Disorder Scale (7 Item) | Baseline to Week 12
  Secondary Mood outcome: self-reported questionnaire to measure the severity of anxiety. Questionnaire ranges 0-24, higher scores indicates greater anxiety state.
PROMIS Applied Cognition Abilities Short | Baseline to Week 12
  Secondary Cognitive outcome:PROMIS (Patient reported outcome measurement information system) is a self-reported questionnaire to measure mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions, ranges from 0-32 , where higher scores indicate improvement.
Attentional Control Scale | Baseline to Week 12
  Secondary Cognitive outcome: The Attentional Control Scale (ACS) is a self-report questionnaire that has been developed to measure individual differences in attentional control. These findings are discussed in relation to previous studies on attentional and executive control in anxiety and depression. Higher scores indicative of better attentional control.
Monetary Incentive Delay Task | Baseline to Week12
  Secondary cognitive outcome. This task assesses neural response during reward anticipation and receipt.
  On each trial, participants are presented with a cue indicating that trial's reward value ($0, $1, $2, or $4). After the cue, a delay period ensues as the participant waits for the target. Participants press a button as quickly as possible when the target is visible. A feedback screen then appears indicating the outcome ("Hit!" or "Miss!") for each trial, with a brief interval before the next trial. Target duration is continually adjusted during the session based on individual performance to keep success rate at 60%. Participants will complete trials over 15 minutes.
Probabilistic Selection Task | Baseline and at week 12
  Secondary cognitive outcome to assess brain's reward system.Participants are instructed to choose between abstract stimuli via key press. The task is composed of two phases. During the first phase, subjects learn to associate 6 abstract visual stimuli with different reward probabilities. In phase 1, the various stimuli are always presented in pairs, where the sum of the two reward probabilities associated with each stimuli equal 100%. Participants learn that for each pair, choosing one stimuli over the other results in more reward. The subject is tested on this association in phase two. During phase two, the subject must decide between novel combinations of stimuli. Each stimuli is presented with the remaining four stimuli that it was not paired with in phase 1. Participants are instructed to win as many rewards as possible

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will include clinical and cognitive, data from older depressed subjects. The final dataset will include clinical information about subject psychiatric diagnoses, psychiatric and medical history, cognitive data, and response to transdermal nicotine. We will share data via the National Institute for Mental Health Data Archive (NDA). NDA provides a secure platform for data-sharing allowing for communication of research data, tools, and supporting documents. As required by NDA, we will obtain a Global Unique Identifier (GUID) for each participant. We will additionally follow NDA requirements to certify and review data, as well as timeline requirements for data submission and data sharing. Sharing of neuroimaging data will also be facilitated by an XNAT system (xnat.org). XNAT is an open-source informatics software platform that assists in the management and archiving of imaging data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared according to policies from the NDA (NIMH Data Archive). Descriptive data, outcome measures and analyzed data will be shared will be shared within 4 months of when a publication is accepted. Study data will be shared through the NDA indefinitely.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Gandelman JA, Kang H, Antal A, Albert K, Boyd BD, Conley AC, Newhouse P, Taylor WD. Transdermal Nicotine for the Treatment of Mood and Cognitive Symptoms in Nonsmokers With Late-Life Depression. J Clin Psychiatry. 2018 Aug 28;79(5):18m12137. doi: 10.4088/JCP.18m12137. PMID 30192444
- [Background] Sutherland MT, Ray KL, Riedel MC, Yanes JA, Stein EA, Laird AR. Neurobiological impact of nicotinic acetylcholine receptor agonists: an activation likelihood estimation meta-analysis of pharmacologic neuroimaging studies. Biol Psychiatry. 2015 Nov 15;78(10):711-20. doi: 10.1016/j.biopsych.2014.12.021. Epub 2015 Jan 7. PMID 25662104
- [Background] Gandelman JA, Newhouse P, Taylor WD. Nicotine and networks: Potential for enhancement of mood and cognition in late-life depression. Neurosci Biobehav Rev. 2018 Jan;84:289-298. doi: 10.1016/j.neubiorev.2017.08.018. Epub 2017 Aug 30. PMID 28859996
- [Background] Aizenstein HJ, Butters MA, Wu M, Mazurkewicz LM, Stenger VA, Gianaros PJ, Becker JT, Reynolds CF 3rd, Carter CS. Altered functioning of the executive control circuit in late-life depression: episodic and persistent phenomena. Am J Geriatr Psychiatry. 2009 Jan;17(1):30-42. doi: 10.1097/JGP.0b013e31817b60af. PMID 19001356
- [Background] Alexopoulos GS, Hoptman MJ, Kanellopoulos D, Murphy CF, Lim KO, Gunning FM. Functional connectivity in the cognitive control network and the default mode network in late-life depression. J Affect Disord. 2012 Jun;139(1):56-65. doi: 10.1016/j.jad.2011.12.002. Epub 2012 Mar 15. PMID 22425432